CLINICAL TRIAL: NCT00930475
Title: Everolimus (RAD001) in Combination With Intravenous Carboplatin in Taxane- and Anthracycline-pretreated Patients With Progressive Metastatic Breast Cancer
Brief Title: Everolimus (RAD001) and Carboplatin in Pretreated Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: KKS Netzwerk (Network); Novartis Pharmaceuticals (Industry)
Responsible Party: Dr. Jan Eucker, Charite University medicine, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001JDE15T
Record Dates: First submitted 2009-06-18; First posted 2009-06-30 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RAD001 (Everolimus) in combination with carboplatin — phase I: dose levels: 2,5 mg, 5 mg, 7,5 mg and 10mg daily in combination with carboplatin AUC2 weekly until progress
Drug: RAD001 (Everolimus) in combination with carboplatin — phase 2: 10mg RAD001 in combination with carboplatin

SUMMARY:
This is an open-label, mono-center phase I/II study designed to determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of RAD001 in combination with carboplatin in taxane- and anthracycline-pretreated patients with progressive metastatic breast cancer. Additionally, the study is designed to characterize the safety, the tolerability and efficacy of this study.

DETAILED DESCRIPTION:
During the phase I part the study will include at least 3 patients at each dose-level until MTD is reached. Each cohort will consist of newly enrolled patients. Intra-patient dose escalation is not permitted. Once MTD is reached a total of 6 patients will be treated at MTD (phase I). For the phase II the minimax two-stage design will be applied. After testing the drug on 16 patients in the first stage of phase II, the trial will be terminated if 1 or fewer respond (SD, PR, CR). If the trial goes on to the second stage, a total of 34 patients will be studied during the phase II part.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients
* at least two prior chemotherapies due to metastatic or inoperable breast cancer
* Karnofsky performance status of at least 60%
* pretreatment with at least one taxane and one anthracycline

Exclusion Criteria:

* previous treatment with mTOR-inhibitors, carboplatin, cisplatin or oxaliplatin
* inadequate organ function including bone marrow function
* bleeding tumours
* known uncontrolled metastases in CNS or carcinomatous meningosis
* patients who have been treated during the last five days with inhibitors or inducers of CYP3A
* serious pulmonary, neurological, endocrinological or other disorders interfering with this study medication, especially patients with known lung fibrosis, emphysema or severe COPD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: dose limiting toxicity | after three weeks
Phase II: response rate | every six weeks

SECONDARY OUTCOMES:
Phase I: adverse events | after three weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité, university medicine, Berlin, CCM, Berlin, State of Berlin, Germany